CLINICAL TRIAL: NCT04716205
Title: Effects of Mulligan's Bent Leg Raise Technique on Hamstring Flexibility and Lumber Spine Mobility in Healthy Females
Brief Title: Mulligan's Bent Leg Raise Technique in Healthy Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REC/LHR/20/1042/Afia Irfan
Record Dates: First submitted 2021-01-19; First posted 2021-01-20 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Hamstring Contractures
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan's bent leg raise Technique (Experimental): Mulligan's bent leg raise Technique and Static Stretching
  Interventions: Other: Mulligan Bent Leg Raise Technique; Other: Static Stretching
- Static stretching (Active Comparator): Static Stretching
  Interventions: Other: Static Stretching

INTERVENTIONS:
Other: Mulligan Bent Leg Raise Technique — Participant will be in supine lying on a high couch with the resting on the shoulder. A distraction (longitudinal traction force along the long axis of femur) will be investigator in walk stand position lateral to the leg, which to be stretch. Hip and Knee of the side to be stretch will bent at 90˚- 90 ˚. Participant's flexed knee will be placed over the shoulder, the popliteal fossa of the knee applied at the lower end of femur and the participant will ask to push the shoulder with his or her leg followed by voluntary relaxation.The traction will maintained throughout the technique.
  Arms: Mulligan's bent leg raise Technique
Other: Static Stretching — It will be given in supine position by performing passive SLR and end range will hold in 30sec.

SUMMARY:
To determine the effects of mulligan's bent leg raise technique on hamstring flexibility and lumber spine mobility in healthy females

DETAILED DESCRIPTION:
Flexibility is a pivotal constituent of the physical fitness and held as an integral aspect that capacitate the person to move smoothly and safely. Although the flexibility of all the muscles of the body is essential for normal human function, the flexibility of hamstring muscle is much emphasized. Investigations suggest adequate flexibility of the Hamstring muscles is compulsory for a healthy lower back. Lack of hamstring muscles extensibility conditions a decrease of pelvic mobility. This invariably leads to biomechanical changes in the pressure distribution of the spine and consequent spinal disorders.

This study will be a randomized control trial and will be conducted in health sciences collage in Bahawalpur. The study will be completed within the time duration of six months. Convenient sampling technique will be used to collect the data. The sample size of 48 patients will be taken in this study to find the Effects of Mulligan's bent leg raise technique on hamstring flexibility and lumber spine mobility in healthy females. Patient will be divided into two groups. Static Stretching will be given to both group as a baseline treatment. (Group A will be treated with Mulligan's bent leg raise techniques and static stretching Group B will be treated with static stretching only. Participants will be assessed for hamstring tightness with Active Knee Extension Test (AKET) and readings will be noted and lumbar mobility will be assess using Modified Schober Test (MMST). Assessments will be done at baseline and post intervention on 5th and 10th day. Intervention will be given 5 days per week for two weeks. Data will be analyzed on SPSS 25.

ELIGIBILITY:
Inclusion Criteria:

* Only healthy females will be included.
* Age 18-24 years.
* BMI normal
* Hamstring muscle tightness -90-90 hip active knee extension test positive (AKET).

Exclusion Criteria:

* Any traumatic and infectious condition involving lower limb.
* Pathologies and deformities related to knee and hip joint.
* Any neurological symptoms affecting the lower limbs.
* Subjects performing regular exercises or stretching.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — * Only healthy females will be included.
  * Age 18-24 years.
  * BMI normal
Enrollment: 44 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Active Knee Extension Test (AKET) | 10 days
  The subject lies supine on a firm table with their head back and arms folded across the chest.
  The hip is passively flexed until the thigh is vertical - use the spirit level to measure the position of the thigh.
  The opposite leg is placed in a fully extended position on the table.
Modified Schobber's Test | 10 days
  The validity of the modified-modified Schober test is moderate (r=0.67) with an excellent interclass (r=0.91) and intraclass (r=95) reliability

CONTACTS AND LOCATIONS:
Overall Officials: Saima Zahid, PhD*, Principal Investigator — Riphah International University
Locations (1):
- king's Rehab center at king's college of Health sciences, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kapadia PD, Meshram VKJI. A comparative study on immediate effects of traction straight leg and bent leg raise on hamstring muscle flexibility in normal individuals. 2019;5(4):274-8.
- [Background] Singh S, Grover V, Singh SJIJoHS, Research. Effect of Neural Mobilization and PNF Stretching on Hamstring Flexibility in working women. 2015;5(8):361-8.
- [Background] Chintamani R, Metgud S, Heggannavar A. Short Term Effects of Instrument Assisted Soft Tissue Mobilisation Technique Versus Mulligan's Bent Leg Raise Technique in Asymptomatic Subjects with Hamstring Tightness-A Randomised Clinical Trial.9(10):50-64.
- [Background] Phadnis T, Bhave SJPR. Comparative Study of Mulligan Bent Leg Raise vs. Hold Relax Proprioceptive Neuromuscular Facilitation on Hamstring Tightness in High School Student. 2018;3(156):2573-0312.1000156
- [Background] Shinde SV, Kanase SBJIJoD, Sciences M. Effect of mulligan bent leg raise versus neural mobilization on hamstring tightness in college students. 2017;16(3):59-63.
- [Background] Dr. Sejal Sathe1 DGMA. To compare the effectiveness of mulligan's bent leg raise and traction straight leg raise on hamstring flexibility in young individuals International Journal of Yoga, Physiotherapy and Physical Education May 2018;Volume 3(Issue 3):Page No. 30-3
- [Background] Khatri S, Yeole U, Kurle S. Effects of various mulligan technique on hamstring muscle imbalance and lumbar spine mobility in marathon runners: A randomized control trial. 2018;5(6):3-6.
- [Background] Yildirim MS, Ozyurek S, Tosun O, Uzer S, Gelecek N. Comparison of effects of static, proprioceptive neuromuscular facilitation and Mulligan stretching on hip flexion range of motion: a randomized controlled trial. Biol Sport. 2016 Mar;33(1):89-94. doi: 10.5604/20831862.1194126. Epub 2016 Feb 8. PMID 26929476
- [Background] Pourahmadi MR, Mohsenifar H, Dariush M, Aftabi A, Amiri A. Effectiveness of mobilization with movement (Mulligan concept techniques) on low back pain: a systematic review. Clin Rehabil. 2018 Oct;32(10):1289-1298. doi: 10.1177/0269215518778321. Epub 2018 May 30. PMID 29843520
- [Background] Tambekar N, Sabnis S, Phadke A, Bedekar N. Effect of Butler's neural tissue mobilization and Mulligan's bent leg raise on pain and straight leg raise in patients of low back ache. J Bodyw Mov Ther. 2016 Apr;20(2):280-5. doi: 10.1016/j.jbmt.2015.08.003. Epub 2015 Aug 14. PMID 27210844
- [Background] 13. Choi Y-j, Sim H-p, Lee J-yJTJoKAoOMPT. The Comparison of Effects Mulligan's Technique Applied to Shortened Hamstring. 2018;24(1):7-14.